CLINICAL TRIAL: NCT03134196
Title: Long-term Suppressive Valacyclovir Treatment for Herpes Zoster Ophthalmicus
Brief Title: Zoster Eye Disease Study
Acronym: ZEDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-00463; 1U10EY026869 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Herpes Zoster Ophthalmicus
Keywords: Herpes Zoster Ophthalmicus; Zoster Eye Disease Study; Varicella Zoster Virus; Zoster; Shingles
MeSH Terms: conditions — Herpes Zoster Ophthalmicus; Chickenpox; Herpes Zoster | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Encapsulated masked placebo
  Interventions: Drug: Masked Placebo
- Masked Oral Valacyclovir 1000 mg daily (Active Comparator): Valacyclovir, 500 mg, oral pill, two 500mg pills daily
  Interventions: Drug: Masked Oral Valacyclovir

INTERVENTIONS:
Drug: Masked Placebo — Oral Placebo
  Arms: Placebo
Drug: Masked Oral Valacyclovir — Oral Valacyclovir 1000 mg/day
  Other Names: Valtrex
  Arms: Masked Oral Valacyclovir 1000 mg daily

SUMMARY:
This is a multi-center, randomized, double-masked, placebo-controlled clinical trial of suppressive valacyclovir for one year in immunocompetent study participants with an episode of dendriform epithelial keratitis, stromal keratitis, endothelial keratitis, and/or iritis due to Herpes Zoster Ophthalmicus (HZO) in the year prior to enrollment.

DETAILED DESCRIPTION:
The objective of the Zoster Eye Disease Study (ZEDS) is to determine whether prolonged suppressive oral antiviral treatment with valacyclovir reduces complications of Herpes Zoster Ophthalmicus (HZO), thereby improving clinical outcomes in this common and potentially vision- and life-threatening disease. There are 1,000,000 new cases of Herpes Zoster (HZ) per year in the USA, with 10-20% being HZO.

Specific Aims

Primary Aim: The primary aim of this double-masked, placebo controlled multicenter randomized clinical trial will test the hypothesis that suppressive antiviral treatment for 12 months with oral valacyclovir 1000 mg daily reduces the rate of new or worsening dendriform epithelial keratitis, stromal keratitis, endothelial keratitis or iritis compared to placebo, at 12 months as the primary endpoint, and at 18 months including 6 months of follow-up after treatment, as a secondary endpoint, in patients with HZO who have had an episode of one of these disease manifestations during the year prior to enrollment.

Secondary Aim: The second aim is to test the hypothesis that suppressive treatment for 12 months with oral valacyclovir 1000 mg daily reduces the severity and duration of postherpetic neuralgia (PHN), compared to placebo, at 12 months and at 18 months as secondary endpoints, in similar patients with HZO. PHN is a debilitating chronic pain syndrome that negatively impacts quality of life, especially in elderly patients.

The study will enroll immunocompetent patients age 18 years and older who have HZO diagnosed at variable times in the past, with these types of active anterior segment ocular segment disease within the past year. Eligible patients will be randomized in a 1:1 ratio to long-term suppressive treatment with oral valacyclovir 1000 mg daily or placebo for 12 months, plus usual ophthalmic care, and followed every 3 months for a total of 18 months, to determine outcomes of new or worsening dendriform epithelial keratitis, stromal keratitis, endothelial keratitis or iritis and/or severity and duration of PHN during 12 months of treatment and for 6 months following treatment discontinuation. The results with regard to PHN may be applicable to HZ in other locations. If suppressive valacyclovir treatment is determined to be effective, the potentially devastating disease burden of HZO and HZ may be reduced for patients, as well as the annual costs to society, estimated in the USA to be one billion dollars.

ELIGIBILITY:
PARTICIPANT INCLUSION CRITERIA

To be eligible for study participation, an individual must meet all of the following criteria:

1. Ability to understand, and willingness and ability to read and sign, the informed consent form.
2. Ability to understand and follow instructions and study procedures.
3. Willingness to comply with all study procedures and be available for the duration of the study.
4. Ability to take oral medication, and are willing to adhere to study medication regimen.
5. Age 18 years or older.
6. Diagnosed with HZO in one eye based on both of these criteria:

   1. History of characteristic unilateral, usually vesicular, HZO rash in the dermatomal distribution of cranial nerve V1 or V2.
   2. Medical record documentation of an episode of active dendriform epithelial keratitis, stromal keratitis, endothelial keratitis, and/or iritis due to HZO within the preceding year. This episode of active anterior segment ocular disease may be due to HZO of recent onset (within the preceding 6 months); or chronic HZO (with onset six or more months ago); may be new, worsening, or recurrent disease after a period of inactivity; and may occur after medication was reduced.

   i. Study participants with chronic HZO must be on a stable treatment regimen and off antivirals for at least 30 days before enrollment. Study participants with chronic HZO who do not meet this criterion may be rescreened, if they are able to meet this criterion within 3 months after the study visit. This is not a requirement for study participants with recent onset HZO, who may be enrolled at any time, preferably after completing recommended acute antiviral treatment, if prescribed, is completed. They can be on variable dose of steroids, and only need to be off oral and topical antivirals by the enrollment visit.
7. For females with reproductive potential, willingness to use highly effective contraception (e.g., hormonal contraception, barrier contraception, intrauterine device, or abstinence).

PARTICIPANT EXCLUSION CRITERIA

An individual who meets any of the following criteria will be excluded from participation in this study:

1. History of immunocompromised status as defined by current CDC contraindications for the vaccine against zoster (44).

   1. Study participants who are diagnosed with leukemia, lymphomas or other malignant neoplasms affecting bone marrow or lymphatic system, unless leukemia in remission and off chemotherapy for at least 3 months.
   2. Study participants who are diagnosed with Acquired Immune Deficiency Syndrome (AIDS) or presents with other clinical manifestations of Human Immunodeficiency virus (HIV) including CD4 count of ≤ 200 cells/ml.
   3. Study participants on immunosuppressive therapy including:

   i. High-dose corticosteroids (greater than equivalent of prednisone 20 mg/day within 1 month) ii. Chemotherapy, other than low dose used for treatment of immune-mediated diseases within 3 months iii. Study participants receiving recombinant human immune mediators and immune modulators, especially antitumor necrosis agents, within 1 month prior to enrollment d. Study participants with unspecified cellular immunodeficiency. e. Study participants with history of hematopoietic stem cell transplantation.
2. Medical history of a systemic disease and thought likely to meet one of the exclusion criteria listed in exclusion criterion #1 during the 18-month study period.
3. Renal insufficiency:

   1. Requires dialysis or has history of renal transplant or
   2. eGFR less than 45, determined within 3 months days preceding enrollment.
4. Allergy or adverse reaction to valacyclovir or acyclovir.
5. History of vaccination against zoster within one month prior to enrollment. Study participants who meet this exclusion criterion may be may be screened and enrollment delayed until eligible within 3 months. If the study participant receives the Herpes Zoster Subunit vaccine (Recombinant Zoster Vaccine (RZV), Shingrix), rescreening should take place one month after the second required dose of the vaccine.
6. Keratorefractive surgery, other than limbal relaxing incisions or astigmatic keratotomies at the time of cataract surgery, within 5 years of enrollment, or keratoplasty of the involved eye with zoster.
7. On systemic antivirals with activity against herpes within the past 30 days, including acyclovir, valacyclovir, or famciclovir, for any reason except for treatment of recent onset HZO, including investigational drug trial.
8. History of another condition that may require treatment with one of these three antivirals listed above in exclusion criterion #7, during the course of the study; study participants who require chronic suppressive antiviral treatment with these medications will be excluded.
9. Sexually active women who are pregnant, nursing, or in their reproductive years who do not agree to use contraception during the 1-year treatment period.
10. Incarceration
11. Any condition or circumstance that in the opinion of the study investigator, would place the study participant in increased risk or affect his/her full compliance or completion of the study.
12. Participation in a clinical study testing a drug, biologic, device or other intervention within the last 30 days from enrollment visit. Study participants who meet this criterion may be rescreened.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Cohen, MD, Study Chair — NYU Langone Health
Locations (78):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Eye Institute, Loma Linda, California
  - Jules Stein Eye Clinic - UCLA, Los Angeles, California
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - UCSF- Francis I. Proctor Foundation, San Francisco, California
  - Pacific Eye Surgeons, Inc., San Luis Obispo, California
  - University of Colorado, Aurora, Colorado
  - Colorado Cornea Consultants P.C., Littleton, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Delray Eye Associates, PA, Delray Beach, Florida
  - University of Florida, Gainesville, Florida
  - Florida Eye Specialists, Jacksonville, Florida
  - University of Miami - Bascom Palmer Eye Institute, Miami, Florida
  - Eye Consultants of Atlanta, PC, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - NorthShore University Health System, Glenview, Illinois
  - Case Western Reserve University, Cleveland, Indiana
  - Indiana University - Glick Eye Institute, Indianapolis, Indiana
  - University of Kansas Medical Center, Prairie Village, Kansas
  - University of Kentucky, Lexington, Kentucky
  - LSU Health Science Center, New Orleans, Louisiana
  - Shreveport Eye Clinic, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - The Krieger Eye Institute, Baltimore, Maryland
  - Wilmer Eye Institute John Hopkins, Bethesda, Maryland
  - Crossroads Eye Physician, Owings Mills, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Medical Center, Peabody, Massachusetts
  - Eye Health Services, Weymouth, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Verdier Eye Center, Grand Rapids, Michigan
  - Northwest Eye Clinic, Golden Valley, Minnesota
  - Jennifer Burdick, Minnetonka, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Opthalmology, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - EyeCare MD of NJ, Morristown, New Jersey
  - Albany Stratton VA Medical Center, Albany, New York
  - Finger Lakes Ophthalmology /The Eye Care Center, Canandaigua, New York
  - Stony Brook Ophthalmology, East Setauket, New York
  - Northwell Health, Great Neck, New York
  - New York Eye and Ear Infirmary, New York, New York
  - NYU Langone Health, New York, New York
  - Weill Cornell Ophthalmology, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Devers Eye Institute, Portland, Oregon
  - Casey Eye Institute - Oregon Health and Science University, Portland, Oregon
  - Vantage Eye Care Center, LLC, Bala-Cynwyd, Pennsylvania
  - Geisinger Eye Clinic, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Corneal Associates at Wills Eye Hospital, Philadelphia, Pennsylvania
  - University of Tennessee - Hamilton Eye Institute, Memphis, Tennessee
  - Cornea and Cataract Consultants of Nashville, Nashville, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Cornea Associates of Texas, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas
  - Cornea Consultants of Texas, Fort Worth, Texas
  - Alkek Eye Center - Baylor College of Medicine, Houston, Texas
  - R and R Eye Research, LLC, San Antonio, Texas
  - University of Utah - Moran Eye Center, Salt Lake City, Utah
  - Virginia Eye Institute, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - NY Eye Surgeons, Seattle, Washington
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (7):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of British Columbia/Vancouver General Hospital Eye Care Centre, Vancouver, British Columbia
  - Kingston Health Sciences Centre-HDH Site and Queen's University, Kingston, Ontario
  - Prism Eye Institute, Oakville, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - The Research Institute of the McGill University Health Centre/McGill Academic Eye Centre, Montreal, Quebec
  - Clinique Axe Visuel, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Warner DB, Jeng BH, Kim J, Liu M, Troxel AB, Hochman JS, Baratz KH, Mian SI, Choulakian MY, Meyer JJ, Lu Y, Twi-Yeboah A, Lee TF, Lopez-Jimenez C, Laury SC, Cohen EJ; ZEDS Trial Research Group. Low-Dose Valacyclovir for Postherpetic Neuralgia in the Zoster Eye Disease Study: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 Apr 1;143(4):277-285. doi: 10.1001/jamaophthalmol.2024.6113. PMID 40048191
- [Derived] Cohen EJ, Troxel AB, Liu M, Hochman JS, Baratz KH, Mian SI, Choulakian MY, Warner DB, Lu Y, Twi-Yeboah A, Lee TF, Kim J, Lopez-Jimenez C, Laury SC, Jeng BH; ZEDS Trial Research Group. Low-Dose Valacyclovir in Herpes Zoster Ophthalmicus: The Zoster Eye Disease Randomized Clinical Trial. JAMA Ophthalmol. 2025 Apr 1;143(4):269-276. doi: 10.1001/jamaophthalmol.2024.6114. PMID 40048183
- [Derived] Prescott CR, Cohen EJ, Hochman JS, Troxel AB, Lu Y, Twi-Yeboah A, Jimenez CL, Mian SI, Mazen CY, Warner DB, Baratz KH, Jeng BH; ZEDS Trial Research Group. Baseline Participant Characteristics at Enrollment in the Zoster Eye Disease Study. Cornea. 2024 Dec 1;43(12):1473-1480. doi: 10.1097/ICO.0000000000003497. PMID 38411973
- [Derived] Cohen EJ, Hochman JS, Troxel AB, Colby KA, Jeng BH; ZEDS Trial Research Group. Zoster Eye Disease Study: Rationale and Design. Cornea. 2022 May 1;41(5):562-571. doi: 10.1097/ICO.0000000000002743. PMID 35090154
- See also: Study website — http://med.nyu.edu/research/zoster-eye-disease-study/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Started | 261 | 266
Completed | 223 | 237
Not Completed | 38 | 29
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 13 | 15
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 19 | 12
Not completed — Site Unable to Contact Participant | 2 | 0
Not completed — Site Closed Scheduling Conflict | 1 | 0
Not completed — Scheduling Conflict | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants were included in the data analysis, not just participants who completed the study. Data were analyzed by intention-to-treat.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily | Total
Number analyzed (Participants) | 261 | 266 | 527
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [49 to 68] | 58 [49 to 66] | 58 [50 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 131 | 266
  Male | 126 | 135 | 261
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 11 | 26
  Not Hispanic or Latino | 246 | 255 | 501
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 4 | 4
  Asian | 13 | 14 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 7 | 22
  White | 222 | 235 | 457
  More than one race | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 34 | 63
  United States | 224 | 226 | 450
  New Zealand | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the First Occurrence of New or Worsening Stromal Keratitis Without Ulceration (SK), Endothelial Keratitis (EK), Iritis (IR), Dendriform Epithelial Keratitis (DEK), or Stromal Keratitis With Ulceration (SKU)
Description: The number of participants with the first confirmed endpoint (new or worsening SK, EK, IR, DEK or SKU associated with pre-specified definitions of these disease manifestations and associated treatment requirements within 12 months in study participants assigned to valacyclovir compared to placebo. Diagnostic criteria were defined using the classification for SK, EK, SKU, and DEK caused by Herpes Simplex Virus (HSV) and standardization of uveitis nomenclature (SUN) for IR. A substantial increase in topical steroid treatment, defined as starting, shifting from a lower to higher potency steroid, or doubling frequency of steroid at one visit (new) or gradually within 3 months (worsening) was required for SK, EK, IR, and SKU.
Time Frame: Month 12
Population: Data were analyzed by intention-to-treat. Treatment requirements for endpoints were revised on January 6, 2020 to allow a recent reduction in steroids for SK, EK, IR, and SKU as the estimated endpoint rate assumed this, and applied retroactively to all endpoints without any knowledge of study outcome data by treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Participants | 86 | 75
Statistical Analysis 1: Comparison: Masked Oral Valacyclovir 1000 mg Daily; Test type: Superiority; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.5 to 1.06], Standard Deviation .11

2. Secondary Outcome: Number of Participants With Persistent Treatment Benefit at 18 Months, 6 Months After Cessation of Treatment
Description: A secondary endpoint, at 18 months, assessed whether the treatment effect persisted 6 months after treatment. Diagnostic criteria were defined using the classification for SK, EK, SKU, and DEK caused by HSV and standardization of uveitis nomenclature (SUN) for IR. A substantial increase in topical steroid treatment, defined as starting, shifting from a lower to higher potency steroid, or doubling frequency of steroid at one visit (new) or gradually within 3 months (worsening) was required for SK, EK, IR, and SKU.
Time Frame: Month 18 (6 months post treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Participants | 104 | 87
Statistical Analysis 1: Comparison: Masked Oral Valacyclovir 1000 mg Daily; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.56 to 0.99], Standard Deviation .04

3. Secondary Outcome: Number of Postherpetic Neuralgia (PHN) Episodes
Description: PHN was defined by a Zoster Brief Pain Inventory (ZBPI) score of ≥ 3 (the level at which pain interferes with normal activities), persisting, occurring, or reoccurring 3 or more months after the onset of Herpes Zoster Ophthalmicus (HZO).
Time Frame: Month 12
Population: Data were analyzed by intention-to-treat.
Measure: Number; unit: Number of PHN episodes
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Number of PHN episodes | 24 | 25

4. Secondary Outcome: Number of Postherpetic Neuralgia (PHN) Episodes
Description: PHN was defined by a ZBPI score of ≥ 3 (the level at which pain interferes with normal activities), persisting, occurring, or reoccurring 3 or more months after the onset of HZO
Time Frame: Month 18 (6 months post treatment)
Population: Data were analyzed by intention-to-treat.
Measure: Number; unit: Number of PHN episodes
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Number of PHN episodes | 20 | 16

5. Secondary Outcome: Average Duration of Postherpetic Neuralgia (PHN) Pain
Description: The duration of pain after zoster is obtained at every visit when they reported pain. Outcome measure was obtained using the Zoster Brief Pain Inventory (ZBPI) score of worst pain in last 24 hours of 3/10 (the level at which pain interferes with normal activities) or more occurring 3 or more months after HZO onset was used to determine the prevalence, severity and duration of PHN.
Time Frame: Month 24 (12 months post-treatment)
Population: Data were analyzed by intention-to-treat.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Months | 14.3 [10.8 to 17.8] | 13.6 [10.7 to 16.4]

6. Secondary Outcome: Average Duration of Postherpetic Neuralgia (PHN) Pain
Description: as for outcome 5
Time Frame: Month 30 (18 months post treatment)
Population: Data were analyzed by intention-to-treat.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
Number analyzed (Participants) | 261 | 266
Months | 18.7 [13.6 to 23.7] | 13.6 [11.6 to 15.6]

ADVERSE EVENTS:
Time Frame: 18 months
Description: PI only monitored for SAEs at every follow-up visit. SAEs reviewed by Clinical Monitor.
Arm/Group | Placebo | Masked Oral Valacyclovir 1000 mg Daily
All-Cause Mortality (participants affected / at risk) | 2/261 | 1/266
Serious Adverse Events (participants affected / at risk) | 18/261 | 19/266
Other Adverse Events (participants affected / at risk) | 0/261 | 0/266
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=261) | Masked Oral Valacyclovir 1000 mg Daily (N=266)
Tachy-brady Syndrome (Cardiac disorders) | 1 | 0
Unstable Angina (Cardiac disorders) | 0 | 1
Heart Attack (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Left Main Coronary Artery Disease (Cardiac disorders) | 1 | 0
Tractional Retinal Detachment with Vitreous Hemorrhage (Eye disorders) | 0 | 1
Severe Gastritis (Gastrointestinal disorders) | 0 | 1
Crohn's Flare (Gastrointestinal disorders) | 0 | 2
Chest Pain (General disorders) | 2 | 0
Pelvic Mass Status Post Pelvic Abscess (General disorders) | 0 | 1
Sepsis with multi-organ failure (General disorders) | 1 | 0
Gallstones (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
COVID-19 Infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinus Infection (Infections and infestations) | 1 | 0
Hospitalization for Viral Respiratory Infection (Infections and infestations) | 0 | 1
Hospitalization for Bronchitis (Infections and infestations) | 0 | 1
Pelvic Abscess complicated by Sepsis (Infections and infestations) | 0 | 1
Postoperative Abdominal Infection (Infections and infestations) | 0 | 1
RSV (Investigations) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fracture of L1 (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intracerebral Hemorrhage (Nervous system disorders) | 1 | 0
Headache (Migraine) (Nervous system disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Nerve blockage secondary to arthritis in the back (Nervous system disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
CT scan shows renal artery stenosis (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COVID-19 Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laparoscopic Appendectomy (Surgical and medical procedures) | 1 | 0
Emergency Open Heart Surgery (Surgical and medical procedures) | 0 | 1
Replacement of Ascending Aortic Aneurysm with Prosthesis (Surgical and medical procedures) | 0 | 1
Ruptured aortic aneurysm (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No Participating Clinical Center (PCC) investigator is permitted to present or publish data obtained during the conduct of this trial without prior approval from the publications committee. PCC investigators must submit a proposal requesting access to trial data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03134196/Prot_SAP_000.pdf